CLINICAL TRIAL: NCT05999149
Title: A Randomized, Open Label, Multicenter Phase III Study of Camrelizumab Plus Chemotherapy in Combination With or Without Famitinib as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (BCTOP-T-N01)
Brief Title: A Study of Camrelizumab Plus Chemotherapy in Combination With or Without Famitinib as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (BCTOP-T-N01)
Acronym: BCTOP-T-N01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCTOP-T-N01
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; Drug Therapy; famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Camrelizumab Plus Chemotherapy and Famitinib
  Interventions: Drug: Camrelizumab Plus Chemotherapy and Famitinib
- Arm B (Active Comparator): Camrelizumab Plus Chemotherapy
  Interventions: Drug: Camrelizumab Plus Chemotherapy

INTERVENTIONS:
Drug: Camrelizumab Plus Chemotherapy and Famitinib — camrelizumab+chemotherapy (Albumin-paclitaxel plus carboplatin)+Famitinib
  Other Names: camrelizumab+chemotherapy+Famitinib
  Arms: Arm A
Drug: Camrelizumab Plus Chemotherapy — Camrelizumab Plus Chemotherapy
  Arms: Arm B

SUMMARY:
This is an open, randomized, controlled, multicenter Phase III clinical study. Eligible subjects were randomly assigned 1:1 to albumin-paclitaxel plus carboplatin and carrilizumab with or without famitinib neoadjuvant therapy. Stratification was performed at randomization according to the following factors: clinical stage of the tumor (stage II; Stage III) and CD8 expression status (IHC ≥10%, < 10%). Subjects who have completed neoadjuvant therapy and are suitable for surgery are required to undergo surgery. Subjects in the experimental group will continue to receive carrilizumab and famitinib until one year from the start of neoadjuvant therapy, and subjects in the control group will continue to receive carrilizumab until one year from the start of neoadjuvant therapy.

Subjects who completed neoadjuvant therapy were required to undergo imaging efficacy evaluation according to RECIST1.1 before surgery; subjects suitable for surgery received surgical treatment, and pathological evaluation of tumor efficacy was performed after surgery.

During the study treatment, if the subjects show disease progression, toxicity intolerance, withdrawal of informed consent, or the investigator determines that medication must be terminated, the study treatment will be terminated, and follow-up will continue, including disease recurrence and metastasis and safety follow-up.

Participants who complete surgical treatment will be followed for at least 2 years for event-free survival (EFS), disease-free survival (DFS), distant metastasis-free survival (DDFS), and safety assessment. Safety data should be collected from the signing of the informed consent until 28 days after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

ECOG Performance Status of 0-1. Early or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression).

Tumor stage: II-III. Adequate hematologic and organ function. Must be willing to use an adequate method of contraception for the course of the study.

Exclusion Criteria:

* Has a history of breast cancer. Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.

Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.

Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4].

Has a diagnosis of immunodeficiency or autoimmune diseases. Has received any form of immunosuppressive therapy within 4 weeks prior to the first dose of study treatment.

Severe pulmonary or cardiac disease. Known active hepatitis C virus, or known active hepatitis B virus. History of organ or bone marrow transplantation. Pregnant or breast-feeding women. Patients who have previously received VEGFR-like small molecule tyrosine kinase inhibitors (such as famitinib, sorafenib, Sunitinib, regorafenib, etc.) (except bevacizumab); Urine routine indicated urinary protein ≥2+ and confirmed urinary protein quantity > 1g at 24h;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to approximately 24 weeks
  the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery

SECONDARY OUTCOMES:
Event-free Survival (EFS) as assessed by Investigator | At least 2 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Disease-free Survival (DFS) as assessed by Investigator | At least 2 years
  DFS is defined as the time from surgery to any of the following events: local or distant recurrence, or death due to any cause.
Distant Disease-free Survival (DDFS) as assessed by Investigator | At least 2 years
  DDFS is defined as the time from surgery to distant recurrence, or death due to any cause.
Objective response rate (ORR) in accordance with RECIST v1.1 | Up to approximately 24 weeks
  Number of responders Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed by MRI.
Number of responders Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed by MRI. | Up to approximately 67 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided